CLINICAL TRIAL: NCT04723732
Title: A Clinical Study Comparing the Antiplaque, Antigingivitis and Anti-inflammatory Effects of Myrrh Mouthwash With Chlorhexidine Mouthwash in a 14-Day Experimental Gingivitis Model
Brief Title: Antiplaque, Antigingivitis and Anti-inflammatory Effects of Myrrh Mouthwash
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, talal zahid, Associate Professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 058-15
Record Dates: First submitted 2020-11-09; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Gingivitis; Dental Plaque
Keywords: gingivitis; herbal; myrrh; myrrha; antigingivitis; antiplaque; IL-1; dental plaque
MeSH Terms: conditions — Gingivitis; Dental Plaque | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Myrrh mouthwash (Experimental): 1% mouthwash of Commiphora myrrha made from resin extract. Participants will use 10 ml of the mouthwash twice daily for 14 days.
  Interventions: Drug: Myrrh mouthwash
- Chlorhexidine Mouthwash (Active Comparator): Commercial 0.2% Chlorhexidine gluconate mouthwash (Avalon Pharma, Riyadh). Participants will use 10 ml of the mouthwash twice daily for 14 days.
  Interventions: Drug: Chlorhexidine mouthwash
- Normal saline (Placebo Comparator): Commercial 0.9% sodium chloride solution (Pharmaceutical solutions industry, Jeddah). Participants will use 10 ml of the mouthwash twice daily for 14 days.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Myrrh mouthwash — 1% mouthwash solution of commiphora myrrha, made from Commiphora Myrrha resin extract.
  Other Names: Commiphora myrrha mouthwash
  Arms: Myrrh mouthwash
Drug: Chlorhexidine mouthwash — 0.2% mouthwash solution of chlorhexidine gluconate.
  Other Names: Chlorhexidine gluconate mouthwash; Avalon Avohex mouthwash
  Arms: Chlorhexidine Mouthwash
Drug: Normal saline — 0.9% solution of sodium chloride, containing 9 g/L Sodium Chloride (154 mEq/L sodium and 154 mEq/L chloride)
  Other Names: Sodium Chloride solution
  Arms: Normal saline

SUMMARY:
Myrrh-based mouthwash has the potential to be a suitable alternative to the gold standard chlorhexidine mouthwash for dental plaque and gingivitis reduction. To date, however, little research has been carried out to determine its true clinical significance on periodontal health. The purpose of this study is to evaluate and compare the efficacy of 1% myrrh mouthwash with commercially available 0.2% chlorhexidine mouthwash in terms of plaque and gingivitis reduction and inflammatory mediator (interleukin-1β) inhibition.

DETAILED DESCRIPTION:
This will be a single-center, triple-blinded, randomized, three-arm parallel, controlled trial in periodontally healthy adult volunteers (no clinical attachment loss and bleeding on probing < 10%). We will include all eligible patients seeking dental treatment at the center after gaining a written informed consent. After the initial dental screening and a session of professional teeth cleaning procedures, participants will be instructed to refrain from regular oral hygiene practices for 2 weeks to develop experimental gingivitis. Participants will then be randomly allocated to one of the three treatment groups [1:1:1] using a simple randomization method (i.e. computer-generated random numbers). They will be instructed to continue refrain from regular oral hygiene practices and use 10 ml of the assigned mouthwash twice daily for 1 minute. Treatment effect will be evaluated by comparing the baseline (day 0) and post-intervention (day 14) values of all clinical parameters (modified gingival index, plaque index, proinflammatory interleukin-1β biomarker, and Gingival Bleeding Index).

ELIGIBILITY:
Inclusion Criteria:

* good periodontal health;
* dentition of ≥20 teeth and a minimum of 5 teeth per quadrant;
* the absence of any systemic illness;
* no history of oral prophylaxis in the past 6 months;
* no relevant medical history that might compromise normal oral hygiene practice.

Exclusion Criteria:

* pocket depth >3 mm
* severe misalignment of teeth;
* the presence of orthodontic appliances;
* intake of antibiotic and/or anti-inflammatory medications within the past 6 months;
* use of tobacco;
* inability of comply with the study's appointment schedule;
* pregnant or breast-feeding mothers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in inflammation on the proinflammatory interleukin (IL)-1β biomarker at Day 14 | Baseline and Day 14
  IL-1β is an important mediator of the inflammatory response. Elevated IL-1β levels have been reported in a number of infectious disease conditions and in noninfectious inflammatory conditions. Human IL-1β ELISA kit by BioVendor was utilized to determine the IL-1β level. Preparation of reagents, execution of test protocol, and calculation of results were done adhering to the manufacturer's Product Data Sheet enclosed with the kit. The absorbance of each strip was read on a spectro-photometer at 450 nm wave length.

SECONDARY OUTCOMES:
Change from Baseline in gingivitis on the 4-point Modified Gingival Index (MGI) at Day 7 and 14 | Baseline, Day 7, and Day 14
  The MGI is a noninvasive visual assessment tool to assess the severity of gingivitis over time. It uses a rating score between 0 (normal gingiva) and 3 (severe inflammation with tendency to spontaneous bleeding). Change = (Day 14 Score - Baseline Score)
Change from Baseline in plaque accumulation on O'leary Plaque Index (PI) at Day 7 and 14 | Baseline, Day 7, and Day 14
  The PI is a validated assessment tool based on recording of the presence of soft debris and mineralized deposits on all 4 surfaces of all teeth. It uses a rating score between 0 (no plaque) and 1 (plaque present at gingival margin). Change = (Day 14 Score - Baseline Score)
Change from Baseline in gingival bleeding on the Gingival Bleeding Index (GBI) at Day 14 | Baseline and Day 14
  The GBI is a reliable indicator of gingival inflammation and periodontal stability. It uses gentle probing of the orifice of the gingival sulcus. The bleeding on probing (BOP) was assessed using a standardized periodontal probe with a 0.6 mm tip and 1 mm marking. A trained examiner measured BOP applying probing forces not exceeding 0.25 N (25 g). A positive finding was recorded if bleeding occured within 10 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Talal Zahid, M.S, Principal Investigator — King Abdulaziz University
Locations (1):
- King Abdul Aziz University, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No